CLINICAL TRIAL: NCT00384982
Title: Myocardial Stem Cell Administration After Acute Myocardial Infarction (MYSTAR) Study: A Multicenter, Randomized Trial Comparing Early and Late Intracoronary or Combined (Intramyocardial and Intracoronary) Administration of Stem Cells
Brief Title: Myocardial Stem Cell Administration After Acute Myocardial Infarction (MYSTAR) Study
Acronym: MYSTAR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Mariann Gyongyosi MD PhD FESC, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Medical University of Vienna
Record Dates: First submitted 2006-10-05; First posted 2006-10-06 (Estimated); Last update posted 2010-01-22 (Estimated); Status verified 2008-08

CONDITIONS: Myocardial Infarction
Keywords: Bone marrow-derived stem cells; Acute myocardial infarction
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A, B, C, D (Experimental): Early or late; percutaneous intracoronary or combined (intramyocardial and intracoronary) administration of BM-MNCs
  Interventions: Procedure: Bone marrow-derived stem cells implantation

INTERVENTIONS:
Procedure: Bone marrow-derived stem cells implantation — percutaneous BM-derived cell therapy
  Other Names: early intracoronary delivery of BM-MNCs; late intracoronary delivery of BM-MNCs; early combined (intramyoc+intracor) delivery of BM-MNCs; late combined (intramyoc+intracor) delivery of BM-MNCs

SUMMARY:
The MYocardial STem cell Administration after acute myocardial infaRction (MYSTAR) study is a multicenter, prospective, randomized, single-blind clinical trial designed to compare the early and late intracoronary or combined (percutaneous intramyocardial and intracoronary) administration of bone marrow-derived stem cells to patients after acute myocardial infarction with reopened infarct-related artery.

DETAILED DESCRIPTION:
Previous data suggest that bone marrow-derived stem cells (BM-SCs) decrease the infarct size and beneficially affect the postinfarction remodeling.

The MYocardial STem cell Administration after acute myocardial infaRction (MYSTAR) study is a multicenter, prospective, randomized, single-blind clinical trial designed to compare the early and late intracoronary or combined (percutaneous intramyocardial and intracoronary) administration of BM-SCs to patients after acute myocardial infarction (AMI) with reopened infarct-related artery.

The primary endpoints are the changes in resting myocardial perfusion defect size and left ventricular ejection fraction (gated SPECT scintigraphy) 3 months after BM-SCs therapy.

The secondary endpoints relate to evaluation of 1) the safety and feasibility of the application modes, 2) the changes in left ventricular wall motion score index (transthoracic echocardiography), 3) myocardial voltage and segmental wall motion (NOGA mapping), 4) left ventricular end-diastolic and end-systolic volumes (contrast ventriculography), and 5) the clinical symptoms (CCS and NYHA) at follow-up.

Patients are randomly assigned into one of four groups, Group A: early treatment (21-42 days after AMI) with intracoronary injection; Group B: early treatment (21-42 days after AMI) with combined (intramyocardial and intracoronary) application; Group C: late treatment (3 months after AMI) with intracoronary delivery; and Group D: late treatment (3 months after AMI) with combined (intramyocardial and intracoronary) administration of BM-SCs. Besides the BM-SCs therapy, the standardized treatment of AMI is applied in all patients.

The MYSTAR trial is the first randomized trial to investigate the effects of the combined (intramyocardial and intracoronary) and the intracoronary mode of delivery of BM-SCs therapy in the early and late periods after AMI.

ELIGIBILITY:
Inclusion Criteria:

* Patient with a definitive AMI not earlier than 21 days and not later than 42 days before randomization (day 0 is the day of infarction)
* Patients with open IRA without significant stenosis and TIMI flow 3, after successful percutaneous coronary intervention (PCI) of the IRA
* Patients with two- or three-vessel disease might be included after adequate PCI if no significant coronary lesion can be seen in the non-infarct-related major vessels at the time of BM-SCs therapy
* A persistent local new wall motion abnormality related to the recent infarct location.
* Preserved myocardial viability, at least in the part of the recent infarction should be demonstrated by a preserved wall thickness and/or hypokinesia determined by transthoracic echocardiography or contrast ventriculography, and preserved tracer uptake determined by early and late resting Thallium myocardial scintigraphy or FDG-PET.
* Global LVEF between 30 and 45%.
* Written informed consent.

Exclusion Criteria:

* Previous heart surgery
* Small posterior or inferior AMI
* Previous MI at the same location
* Regional wall motion abnormality outside the area involved in the index AMI
* Ventricular thrombus
* Severe valvular heart disease
* Severe renal, lung and liver disease
* Disease of the hematopoetic system
* Hemoglobin level below 9 mg%
* The patient cannot follow the study protocol
* NYHA functional class IV at baseline
* Postinfarct angina
* Significant coronary stenosis in the IRA requiring repeated PCI at the time of the planned BM-SCs therapy
* Significant coronary lesion in one or more major coronary vessels, requiring revascularization
* Age lower than 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2005-01; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Changes in resting myocardial perfusion defect size by gated SPECT scintigraphy 3-6 months after the percutaneous intracoronary or combined bone marrow-derived stem cells therapy. | 3-6 month
Changes in global left ventricular ejection fraction by gated SPECT scintigraphy 3-6 months after the percutaneous intracoronary or combined bone marrow-derived stem cells therapy. | 3-6 month

SECONDARY OUTCOMES:
The feasibility of the bone marrow-derived stem cells delivery modes, determined by the rates of acute and subacute complications | in-hospital
Change in the left ventricular wall motion score index, measured by transthoracic echocardiography | 3-6 month
Change in the myocardial voltage as a parameter of myocardial viability obtained by NOGA endocardial mapping, with segmental wall motion expressed by local linear shortening on NOGA mapping | 3-6 month
Change in left ventricular end-diastolic and end-systolic volumes by contrast ventriculography | 3-6 month
Assessment of the clinical symptoms (CCS and NYHA) of the patients | 3, 6 and 12 month
The safety of the bone marrow-derived stem cells delivery modes, expressed as the rates of long-term major adverse cardiac events (MACE: death, target vessel revascularization and non-fatal AMI) | 3, 6 and 12 month

CONTACTS AND LOCATIONS:
Overall Officials: Irene Lang, MD, Study Director — Department of Cardiology, Medical University of Vienna; Dietmar Glogar, MD, Study Chair — Department of Cardiology, Medical University of Vienna; Mariann Gyongyosi, MD, Principal Investigator — Department of Cardiology, Medical University of Vienna
Locations (1):
- Department of Cardiology, Medical University of Vienna, Vienna, Austria